CLINICAL TRIAL: NCT04808895
Title: Multicenter Randomized, Double-blind, Placebo-controlled, Clinical Trial of Acetylsalicylic Acid in the Prevention of Severe SARS-CoV2 Pneumonia in Hospitalised Patients (Asperum)
Brief Title: Acetylsalicylic Acid in the Prevention of Severe SARS-CoV2 Pneumonia in Hospitalised Patients With COVID-19
Acronym: Asperum
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2020-006130-12
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; Thrombosis Pulmonary
Keywords: Acetylsalicylic acid; Heparin; Pulmonary thrombosis; COVID-19; Platelets; Inflammation; Respiratoty failure
MeSH Terms: conditions — COVID-19; Inflammation | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Experimental phase 3 drug trial, randomized 1:1, double-blind, multicentre in patients treated with acetylsalicylic acid vs placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Use of placebo tablets of the same shape, colour of the investigational drug. Identical time and route of administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylsalicylic acid (Active Comparator): Tablets of 100 mg acetylsalicylic acid (one 100 mg daily dose. On the first day a loading dose of 300 mg will be administered)
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator): Tablets of placebo, identical to active comparator (one tablet daily dose. On the first day 3 tablets will be administered)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid — administration of one tablet daily for 15 days. On the first day a loading dose of 300 mg will be administered
  Arms: Acetylsalicylic acid
Drug: Placebo — administration of one tablet daily for 15 days. On the first day 3 tablets will be administered
  Arms: Placebo

SUMMARY:
Inflammatory diseases favour the onset of venous thromboembolic events in hospitalized patients. Thromboprophylaxis with a fixed dose of heparin/low molecular weight heparin (LMWH) is recommended if concomitant inflammatory disease. In severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) pneumonia an inflammation-dependent thrombotic process occurs and platelet activation may promote thrombosis and amplify inflammation, as indicated by previous experimental evidence, and the similarities with atherothrombosis and thrombotic microangiopathies. Antiplatelet agents represent the cornerstone in the prevention and treatment of atherosclerotic arterial thromboembolism, with limited efficacy in the context of venous thromboembolism. The use of acetylsalicylic acid may improve inflammation and respiratory function in humans as indicated by the results of observational studies. There are no validated protocols for thrombosis prevention in Covid-19. There is scientific rationale to consider acetylsalicylic acid for the prevention of thrombosis in the pulmonary circulation and attenuation of inflammation. This is supported by numerous demonstrations of the anti-inflammatory activity of antiplatelet agents and the evidence of improvement in respiratory function both in human and experimental pathology. The hypothesis underlying the present study project is that in Covid-19 platelet activation occurs through an inflammation-dependent mechanism and that early antithrombotic prophylaxis in non-critical patients could reduce the incidence of pulmonary thrombosis and respiratory and multi-organ failure improving clinical outcome in patients with SARS-CoV2 pneumonia. The prevention of thrombogenic platelet activity with acetylsalicylic acid could be superior to fixed dose enoxaparin alone. The proposed treatment is feasible in all coronavirus disease 2019 (COVID-19) patients, regardless of the treatment regimen (antivirals, anti-inflammatory drugs), except for specific contraindications. To this aim, the investigators a randomised, placebo-controlled, double blind, parallel arms study to investigate the potential protection of acetylsalicylic acid towards the progression of lung failure in patients admitted to a medical ward for SARS-CoV-2 pneumonia. A 15-day treatment period is considered. Primary endpoint is the occurrence of one of the following events: admission to an intensive care unit, requirement of mechanical ventilation, PaO2/FiO2 less than 150 mm Hg.

DETAILED DESCRIPTION:
Severe respiratory failure and multi-organ damage in coronavirus disease 2019 (COVID-19) patients have not a unitary pathophysiological interpretation. There is evidence of an association between the clinical entity of the disease and its severity with the plasma levels of D-dimer and inflammatory indexes. On the basis of retrospective investigations there is accumulating evidence of alterations in the haemostatic parameters that with increased D-dimer values, increased coagulation time and platelets may be predictors of worse prognosis. A systematic survey conducted in the coronavirus disease 2019 (COVID-19) Centre of the AOUI Verona, as part of the Database and Study on the role of platelets in the clinical manifestations of COVID-19 (Ethics Committee CESC Verona and Rovigo approved) revealed by means of computerized tomography (CT) angiograph in patients with a persistent respiratory deficit and very high D-dimer values mainly multiple, bilateral vascular occlusions involving the segmental and subsegmental branches of the pulmonary arteries. This finding is suggestive of a frequent and clinically relevant thrombotic process in a appreciable number (approximately 20%) of patients with COVID-19 pneumonia hospitalized in medical wards. It is a well-established clinical notion that acute and chronic inflammatory diseases may favour the onset of venous thromboembolic events in hospitalized patients. Thromboprophylaxis with a fixed dose of heparin/low molecular weight heparin (LMWH) is recommended for medical patient with concomitant neoplasia or inflammatory disease. It is conceivable that under conditions, such as SARS-CoV2 pneumonia, an inflammation-dependent thrombotic process takes place and that platelet activation may play a pathogenic role both in the thrombotic process and in the amplification of the inflammatory process. In fact, there is experimental evidence that platelet activation in inflammation would lead to accelerated coagulation and a thrombotic vascular occlusion, with similarities to what is widely documented in atherothrombosis and thrombotic microangiopathies. The administration of antiplatelet drugs represents the cornerstone for the prevention and treatment of arterial thromboembolism in atherosclerotic disease and has also shown some limited efficacy also in the context of venous and arterial thromboembolism associated with atrial fibrillation. The use of acetylsalicylic acid may improve inflammation and respiratory function in humans as indicated by the results of observational studies. There are currently no validated protocols for thrombosis prevention in the field of pulmonary viral diseases, in particular COVID-19. There is scientific rationale to consider acetylsalicylic acid for the prevention of thrombosis in the pulmonary circulation and attenuation of inflammation. This is supported by numerous demonstrations of the anti-inflammatory activity of antiplatelet agents and the evidence of improvement in respiratory function both in human and experimental pathology. A retrospective observational study showed that patients with COVID-19 pneumonia treated with acetyl salicylic acid had a lower incidence of progression to respiratory failure requiring mechanical ventilation, without evidence of increased incidence of bleeding complications. The hypothesis underlying the present study project is that in Covid-19 platelet activation occurs via an inflammation-dependent mechanism and that early antithrombotic prophylaxis in non-critical patients, like those admitted to medical wards, could reduce the incidence of pulmonary thrombosis as well as respiratory and multi-organ failure, contributing to improve clinical outcome of the patients with pneumonia caused by SARS-CoV2 viruses. The anticoagulant activity exerted by a fixed dose of enoxaparin (4000U/day), recommended in patients with the described clinical features, according to a note of the "Italian Medicines Agency" (AIFA), together with the prevention of thrombogenic activity of platelets by acetylsalicylic acid could prevent aggravation of COVID-19 patients to a greater extent than enoxaparin alone given at the same dose. Early initiation of treatment should mitigate the presentation of pneumonia. The proposed treatment is feasible in all coronavirus disease 2019 (COVID-19) patients, regardless of the treatment regimen (antivirals, anti-inflammatory drugs), except for specific contraindications. To this aim, it was designed a randomised, placebo-controlled, double blind, parallel arms study to investigate the potential protection of acetylsalicylic acid towards the progression of lung failure in patients admitted to a medical ward for SARS-CoV-2 pneumonia. A 15-day treatment period is considered. Primary endpoint is the occurrence of one of the following events: admission to an intensive care unit, requirement of mechanical ventilation, PaO2/FiO2 less than 150 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* in a medical area ward dedicated to Covid-19 patients
* Positivity by RT_PCR of the search for genetic material of SARS-CoV2
* Covid-19 pneumonia with moderate clinical picture based on clinical parameters
* O2 saturation> 94% with maximum FiO2 32%
* Respiratory acts <30 / minute
* age >18 years
* Consent to participate in the study

Exclusion Criteria:

* Any Antithrombotic treatment including acetylsalicylic acid
* Active Bacterial infection
* Active or in maintenance therapy neoplasm
* Inability to provide consent
* Any contraindication to the acetylsalicylic acid use
* Active peptic disease
* Active Major pathological bleeding
* Recent (<30 days) major bleeding
* Recent intracranial bleeding
* Need to use therapeutic doses of oral anticoagulants or heparins
* Need to use combination antiplatelet drugs for clinical indication
* Hypersensitivity to acetylsalicylic acid or to any of the excipients
* Hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs)
* Severe hepatic insufficiency (Child-Pugh class C).
* Severe heart failure (NYHA class 3-4)
* Platelet count less than 150000 / mmc
* Haemostasis alteration (INR> 1.5, APTT> 1.5)
* Plasma fibrinogen <100 mg / dL
* Blood pressure >160/100 mmHg
* Concomitant treatment with serotonin reuptake inhibitors
* Participation in another pharmacological clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of clinical worsening | day 15
  Transfer to ICU
Prevention of lung function worsening | day 15
  PaO2/FiO2 lower than 150 mm Hg
Prevention of death | day 15
  Death for any cause

SECONDARY OUTCOMES:
Change in body temperature | Daily for 15 days
  Body temperature
Change in oxygen saturation | Daily for 15 days
  Oxygen saturation
Change in blood gases | Daily for 15 days
  blood gas analysis
Change in blood cell count | Daily for 15 days
  blood cell count
Change in blood oxygen | Daily for 15 days
  Oxygen administration when O2 saturation <92%
Change in clinical markers of lung function | Daily for 15 days
  PaO2/FiO2; progression of disease at Rx
Change in clinical markers of liver damage | Daily for 15 days
  markers of organ damage (ALT)
Change in clinical markers of hearth damage | Daily for 15 days
  markers of organ damage (troponin)
Change in clinical markers of renal damage | Daily for 15 days
  markers of organ damage (creatinine)
Effects on blood cell count | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers (blood cell count)
Effects on CRP | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers (CRP)
Effects on D-dimer | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers (D-dimer)
Effects on interleukin-1 | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers ( IL-1)
Effects on interleukin-6 | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers (IL-6)
Effects on fibrinogen | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers (fibrinogen)
Effects on plasma albumin | Baseline, day 1, 2, 7 and 15.
  Inflammatory markers (albumin)
Effects on protrombin time | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (prothrombin time)
Effects on activated partial thromboplastin time | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (activated partial thromboplastin time)
Effects on serum thromboxane | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets ( serum TxB2)
Effects on thromboxane metabolite | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (urinary 11-dehydro TXB2)
Effects on platelet count | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (platelet count)
Effects on reticulated platelets | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (reticulated platelets)
Effects on platelet/leukocyte conjugates | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (platelets/leukocytes conjugates)
Effects on plasma P-selectin | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (plasma P-selectin)
Effects on P-selectin expression | Baseline, day 1, 2, 7 and 15.
  platelet and hemostatic markets (platelet expression of P-selectin)
Clincal mixed outcome of lung function, ROX score | Days 7 and 15
  ROX score
Clincal mixed outcome of lung function, SOfa score | Days 7 and 15
  SOfa score
Clincal mixed outcome of lung function, Apache index | Days 7 and 15
  Apache index
Clincal mixed outcome of lung function, need to perform CT scan due to worsening of blood gases | Days 7 and 15
  need to perform CT scan due to worsening of blood gases
Clincal mixed outcome of lung function, need to transfer the patient to ICU | Days 7 and 15
  need to transfer the patient to ICU
Clincal mixed outcome of lung function, need for mechanical ventilation | Days 7 and 15
  need for mechanical ventilation
Clincal mixed outcome of lung function, days without need of mechanical ventilation | Days 7 and 15
  days without need of mechanical ventilation
Clincal mixed outcome of lung function, venous thromboembolism | Days 7 and 15
  venous thromboembolism
Clincal mixed outcome of lung function, pulmonary thrombosis | Days 7 and 15
  pulmonary thrombosis
Clincal mixed outcome of lung function, cardiovascular event | Days 7 and 15
  cardiovascular event
Clincal mixed outcome of lung function, death | Days 7 and 15
  death
Clincal mixed outcome of lung function, multiorgan failure | Days 7 and 15
  multiorgan failure
Clincal mixed outcome of lung function, discharge due to resolution of signs and symptoms | Days 7 and 15
  discharge due to resolution of signs and symptoms
Safety outcomes, Major or clinically relevant bleeding | days 1,2,7 and 15
  Major or clinically relevant bleeding
Safety outcomes, total bleeding based on ISTH bleeding score | days 1,2,7 and 15
  total bleeding based on ISTH bleeding score
Safety outcomes, minor bleeding according to ISTH BS | days 1,2,7 and 15
  minor bleeding according to ISTH BS
Safety outcomes, decrease in platelet count below 100x109/L | days 1,2,7 and 15
  decrease in platelet count below 100x109/L
Safety outcomes, decrease of al least 2 g/dl Hb levels | days 1,2,7 and 15
  decrease of al least 2 g/dl Hb levels
Safety outcomes, need for blood transfusion | days 1,2,7 and 15
  need for blood transfusion
Safety outcomes, alterations of clinical or laboratory parameters | days 1,2,7 and 15
  alterations of clinical or laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Minuz, Professor, Study Director — University of Verona, AOUI Verona; Marco Cattaneo, Professor, Study Director — University of Milan; Roberto Leone, Professor, Study Director — Universita di Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

REFERENCES:
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Background] Becattini C, Agnelli G, Schenone A, Eichinger S, Bucherini E, Silingardi M, Bianchi M, Moia M, Ageno W, Vandelli MR, Grandone E, Prandoni P; WARFASA Investigators. Aspirin for preventing the recurrence of venous thromboembolism. N Engl J Med. 2012 May 24;366(21):1959-67. doi: 10.1056/NEJMoa1114238. PMID 22621626
- [Background] Bianconi V, Violi F, Fallarino F, Pignatelli P, Sahebkar A, Pirro M. Is Acetylsalicylic Acid a Safe and Potentially Useful Choice for Adult Patients with COVID-19 ? Drugs. 2020 Sep;80(14):1383-1396. doi: 10.1007/s40265-020-01365-1. PMID 32705604
- [Background] Carestia A, Davis RP, Grosjean H, Lau MW, Jenne CN. Acetylsalicylic acid inhibits intravascular coagulation during Staphylococcus aureus-induced sepsis in mice. Blood. 2020 Apr 9;135(15):1281-1286. doi: 10.1182/blood.2019002783. PMID 31951648
- [Background] Cattaneo M, Bertinato EM, Birocchi S, Brizio C, Malavolta D, Manzoni M, Muscarella G, Orlandi M. Pulmonary Embolism or Pulmonary Thrombosis in COVID-19? Is the Recommendation to Use High-Dose Heparin for Thromboprophylaxis Justified? Thromb Haemost. 2020 Aug;120(8):1230-1232. doi: 10.1055/s-0040-1712097. Epub 2020 Apr 29. No abstract available. PMID 32349132
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Chow JH, Khanna AK, Kethireddy S, Yamane D, Levine A, Jackson AM, McCurdy MT, Tabatabai A, Kumar G, Park P, Benjenk I, Menaker J, Ahmed N, Glidewell E, Presutto E, Cain S, Haridasa N, Field W, Fowler JG, Trinh D, Johnson KN, Kaur A, Lee A, Sebastian K, Ulrich A, Pena S, Carpenter R, Sudhakar S, Uppal P, Fedeles BT, Sachs A, Dahbour L, Teeter W, Tanaka K, Galvagno SM, Herr DL, Scalea TM, Mazzeffi MA. Aspirin Use Is Associated With Decreased Mechanical Ventilation, Intensive Care Unit Admission, and In-Hospital Mortality in Hospitalized Patients With Coronavirus Disease 2019. Anesth Analg. 2021 Apr 1;132(4):930-941. doi: 10.1213/ANE.0000000000005292. PMID 33093359
- [Background] Connors JM, Levy JH. COVID-19 and its implications for thrombosis and anticoagulation. Blood. 2020 Jun 4;135(23):2033-2040. doi: 10.1182/blood.2020006000. PMID 32339221
- [Background] Gu SX, Tyagi T, Jain K, Gu VW, Lee SH, Hwa JM, Kwan JM, Krause DS, Lee AI, Halene S, Martin KA, Chun HJ, Hwa J. Thrombocytopathy and endotheliopathy: crucial contributors to COVID-19 thromboinflammation. Nat Rev Cardiol. 2021 Mar;18(3):194-209. doi: 10.1038/s41569-020-00469-1. Epub 2020 Nov 19. PMID 33214651
- [Background] Jackson SP, Darbousset R, Schoenwaelder SM. Thromboinflammation: challenges of therapeutically targeting coagulation and other host defense mechanisms. Blood. 2019 Feb 28;133(9):906-918. doi: 10.1182/blood-2018-11-882993. Epub 2019 Jan 14. PMID 30642917
- [Background] Hottz ED, Azevedo-Quintanilha IG, Palhinha L, Teixeira L, Barreto EA, Pao CRR, Righy C, Franco S, Souza TML, Kurtz P, Bozza FA, Bozza PT. Platelet activation and platelet-monocyte aggregate formation trigger tissue factor expression in patients with severe COVID-19. Blood. 2020 Sep 10;136(11):1330-1341. doi: 10.1182/blood.2020007252. PMID 32678428
- [Background] Koupenova M, Corkrey HA, Vitseva O, Manni G, Pang CJ, Clancy L, Yao C, Rade J, Levy D, Wang JP, Finberg RW, Kurt-Jones EA, Freedman JE. The role of platelets in mediating a response to human influenza infection. Nat Commun. 2019 Apr 16;10(1):1780. doi: 10.1038/s41467-019-09607-x. PMID 30992428
- [Background] Margraf A, Zarbock A. Platelets in Inflammation and Resolution. J Immunol. 2019 Nov 1;203(9):2357-2367. doi: 10.4049/jimmunol.1900899. PMID 31636134
- [Background] Marongiu F, Mameli A, Grandone E, Barcellona D. Pulmonary Thrombosis: A Clinical Pathological Entity Distinct from Pulmonary Embolism? Semin Thromb Hemost. 2019 Nov;45(8):778-783. doi: 10.1055/s-0039-1696942. Epub 2019 Sep 19. PMID 31537029
- [Background] Middleton EA, He XY, Denorme F, Campbell RA, Ng D, Salvatore SP, Mostyka M, Baxter-Stoltzfus A, Borczuk AC, Loda M, Cody MJ, Manne BK, Portier I, Harris ES, Petrey AC, Beswick EJ, Caulin AF, Iovino A, Abegglen LM, Weyrich AS, Rondina MT, Egeblad M, Schiffman JD, Yost CC. Neutrophil extracellular traps contribute to immunothrombosis in COVID-19 acute respiratory distress syndrome. Blood. 2020 Sep 3;136(10):1169-1179. doi: 10.1182/blood.2020007008. PMID 32597954
- [Background] Minuz P, Mansueto G, Mazzaferri F, Fava C, Dalbeni A, Ambrosetti MC, Sibani M, Tacconelli E. High rate of pulmonary thromboembolism in patients with SARS-CoV-2 pneumonia. Clin Microbiol Infect. 2020 Nov;26(11):1572-1573. doi: 10.1016/j.cmi.2020.06.011. Epub 2020 Jun 18. No abstract available. PMID 32565320
- [Background] Patrono C, Baigent C. Role of aspirin in primary prevention of cardiovascular disease. Nat Rev Cardiol. 2019 Nov;16(11):675-686. doi: 10.1038/s41569-019-0225-y. Epub 2019 Jun 26. PMID 31243390
- [Background] Pulavendran S, Rudd JM, Maram P, Thomas PG, Akhilesh R, Malayer JR, Chow VTK, Teluguakula N. Combination Therapy Targeting Platelet Activation and Virus Replication Protects Mice against Lethal Influenza Pneumonia. Am J Respir Cell Mol Biol. 2019 Dec;61(6):689-701. doi: 10.1165/rcmb.2018-0196OC. PMID 31070937
- [Background] Scavone M, Rizzo J, Femia EA, Podda GM, Bossi E, Caberlon S, Paroni R, Cattaneo M. Patients with Essential Thrombocythemia may be Poor Responders to Enteric-Coated Aspirin, but not to Plain Aspirin. Thromb Haemost. 2020 Oct;120(10):1442-1453. doi: 10.1055/s-0040-1714351. Epub 2020 Jul 27. PMID 32717754
- [Background] Sexton TR, Zhang G, Macaulay TE, Callahan LA, Charnigo R, Vsevolozhskaya OA, Li Z, Smyth S. Ticagrelor Reduces Thromboinflammatory Markers in Patients With Pneumonia. JACC Basic Transl Sci. 2018 Aug 28;3(4):435-449. doi: 10.1016/j.jacbts.2018.05.005. eCollection 2018 Aug. PMID 30175268
- [Background] Simes J, Becattini C, Agnelli G, Eikelboom JW, Kirby AC, Mister R, Prandoni P, Brighton TA; INSPIRE Study Investigators (International Collaboration of Aspirin Trials for Recurrent Venous Thromboembolism). Aspirin for the prevention of recurrent venous thromboembolism: the INSPIRE collaboration. Circulation. 2014 Sep 23;130(13):1062-71. doi: 10.1161/CIRCULATIONAHA.114.008828. Epub 2014 Aug 25. PMID 25156992
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Taus F, Salvagno G, Cane S, Fava C, Mazzaferri F, Carrara E, Petrova V, Barouni RM, Dima F, Dalbeni A, Romano S, Poli G, Benati M, De Nitto S, Mansueto G, Iezzi M, Tacconelli E, Lippi G, Bronte V, Minuz P. Platelets Promote Thromboinflammation in SARS-CoV-2 Pneumonia. Arterioscler Thromb Vasc Biol. 2020 Dec;40(12):2975-2989. doi: 10.1161/ATVBAHA.120.315175. Epub 2020 Oct 14. PMID 33052054
- [Background] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Background] Wichmann D, Sperhake JP, Lutgehetmann M, Steurer S, Edler C, Heinemann A, Heinrich F, Mushumba H, Kniep I, Schroder AS, Burdelski C, de Heer G, Nierhaus A, Frings D, Pfefferle S, Becker H, Bredereke-Wiedling H, de Weerth A, Paschen HR, Sheikhzadeh-Eggers S, Stang A, Schmiedel S, Bokemeyer C, Addo MM, Aepfelbacher M, Puschel K, Kluge S. Autopsy Findings and Venous Thromboembolism in Patients With COVID-19: A Prospective Cohort Study. Ann Intern Med. 2020 Aug 18;173(4):268-277. doi: 10.7326/M20-2003. Epub 2020 May 6. PMID 32374815
- [Background] Yin S, Huang M, Li D, Tang N. Difference of coagulation features between severe pneumonia induced by SARS-CoV2 and non-SARS-CoV2. J Thromb Thrombolysis. 2021 May;51(4):1107-1110. doi: 10.1007/s11239-020-02105-8. PMID 32246317
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818